CLINICAL TRIAL: NCT04775459
Title: Surfactant Replacement Guided by Early Lung Ultrasound Score (LUS) in Preterm Newborns < 33 Weeks With Respiratory Distress Syndrome in the Neonatal Intensive Care Unit of Saint-Etienne.
Brief Title: Surfactant Replacement Guided by Early Lung Ultrasound Score in Preterm Newborns With Respiratory Distress Syndrome
Acronym: ECHOSURF
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN232021/CHUSTE
Record Dates: First submitted 2021-02-25; First posted 2021-03-01 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Preterm Birth
Keywords: Preterm; Lung Ultrasound Score; Surfactant
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Surfactant administration without using score LUS: It is a retrospective cohort : preterm newborns from august 2019 to december 2019 needed a surfactant administration.
  The surfactant was administrated only if the fraction of inspired oxygen (FiO2) >30% among the Guidelines of 2019
  Interventions: Drug: Surfactant administration until 2020
- Surfactant administration using score LUS: It is a prospective cohort : preterm newborns from january 2021 to juin 2020 needed a surfactant administration.
  The surfactant is administrated if FiO2 >30% OR if score LUS >8/18 among the literature
  Interventions: Drug: Surfactant administration since 2021

INTERVENTIONS:
Drug: Surfactant administration until 2020 — Surfactant is administrated if Fi02 >30% among the Guidelines of 2019
  Other Names: No LUS
  Groups: Surfactant administration without using score LUS
Drug: Surfactant administration since 2021 — Surfactant is administrated if Fi02 >30% OR if score LUS >8/18 among the literature
  Other Names: With LUS
  Groups: Surfactant administration using score LUS

SUMMARY:
Lung immaturity is a major issue in neonatal unit.The surfactant administration improves the pulmonary prognosis in premature infants with hyaline membrane disease who escape continuous positive airway pressure (CPAP).

This surfactant had been administered at 5h25min of life in Saint Etienne from 2016 to 2019.

Studies suggest that the earlier the surfactant is administered, the more it can reduce the rate of bronchodysplasia and mortality. And some studies show a pulmonary ultrasound could help to administrate the surfactant earlier This is why a new faster strategy for diagnosing preterms needing surfactant will be usefulness and have been done in Saint-Etienne since 2021 thanks to a ultrasound score (LUS).

DETAILED DESCRIPTION:
This current study analyzes the impact of early Lungs Ultrasounds which use a semi-quantitative assessment : the Lung Ultrasound Score (LUS), in preterms <33 weeks on the time to surfactant administration.

The current hypothesis is that Lung Ultrasound can increase the number of preterms with surfactant replacement within the first 3 hours of life.

This is a prospective, comparative, observational trial between two different cohorts : the last 6 months of 2019 (without Score LUS) versus the first 6 months of 2021 (with Score LUS).

ELIGIBILITY:
Inclusion Criteria:

* newborns <33 weeks old
* born at the Saint Etienne University Hospital
* respiratory distress syndrome

Exclusion Criteria:

* chromosomal abnormality,
* multi-polymalformations syndrome,
* congenital pulmonary disease,
* septic shock,
* congenital lung infection,
* meconium inhalation,
* pneumothorax
* conditions requiring surgery in the first week of life.

Max Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: preterm newborns < 33 weeks with Respiratory Distress Syndrom needed surfactant administration
  Date of birth from 01/08/19 to 31/12/19 and from 01/01/21 to 30/06/21
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
administration time frame (min of life) | day 1
  Time from birth to surfactant administration

SECONDARY OUTCOMES:
FiO2 maximum | Week 1
  Collect in medical record.: the maximal value of FiO2 from birth to one week of life
delay from FiO2 maximum to FiO2 < 21% | Week 4
  Collect in medical record
Ventilation time (day) | Week 4
  Collect in medical record : number of day using a ventilation
Ventilation support | Week 4
  Collect in medical record : using a invasive ou a non invasive ventilation
Bronchodysplasia rate | Week 4
  Collect in medical record.

CONTACTS AND LOCATIONS:
Overall Officials: Aurelie CANTAIS, MD, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- Chu de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No